CLINICAL TRIAL: NCT03222440
Title: A Single Arm Exploratory Study of Radiation Therapy With Anti-PD-1 Antibody SHR-1210 in Treating Patients With Locally Advanced Esophageal Squamous Cell Carcinomas
Brief Title: Combination of Radiotherapy and SHR-1210 to Treat Patients With ESCC
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Tianjin Medical University Cancer Institute and Hospital (Other)
Collaborators: Jiangsu HengRui Medicine Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SHR-1210-RT-ESC-IIT
Record Dates: First submitted 2017-07-13; First posted 2017-07-19 (Actual); Last update posted 2019-12-04 (Actual); Status verified 2019-11

CONDITIONS: Esophageal Cancer
MeSH Terms: conditions — Esophageal Neoplasms | interventions — camrelizumab; spartalizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- SHR-1210+ Radiotherapy (Experimental): Radiotherapy,intensity modulated radiation therapy (IMRT), 54-60 Gy, 1.8-2.0 Gy per fraction ,5 fractions per week, for 6 weeks. Radiation begun the day after the first dose of SHR-1210. SHR-1210 (200mg fixed dose every 2 weeks, one cycle is four weeks, total 8 cycles ) will be administered as an intravenous infusion over 30 minutes.
  Interventions: Drug: SHR-1210

INTERVENTIONS:
Drug: SHR-1210 — SHR-1210 is a humanized anti-PD1 IgG4 monoclonal antibody.
  Other Names: Anti-PD-1 Antibody

SUMMARY:
SHR-1210 is a humanized anti-PD1 IgG4 monoclonal antibody. This is an open-label，single center ，non-randomized ，Single Arm Exploratory Study . This clinical study is an investigator-initiatedclini-cal trial（IIT ）.The objective of this study is to evaluate the efficacy and safety of radiation therapy combined with anti-PD-1 antibody SHR-1210 in patients with Locally Advanced Esophageal Squamous Cell Carcinomas。

ELIGIBILITY:
Inclusion Criteria:

1. age:18-75 years, male or femal.
2. Histologically confirmed primary Squamous Cell Carcinoma of the Esophagus,Local advanced esophageal cancer diagnosed by pathology and imaging,clinical stage T3-4N0M0, T1-4N+M0,Ⅱ-Ⅳa.
3. Pre-treatment evaluation can not tolerate concurrent radiochemotherapy or rejection of the concurrent use of chemotherapy with radiotherapy.
4. Measurable disease based on Response Evaluation Criteria In Solid Tumors (RECIST) 1.1.
5. ECOG 0-1.
6. Adequate organ function.
7. Life expectancy of greater than 6 months.
8. Patient has given written informed consent.

Exclusion Criteria:

1. Patients who have or are currently undergoing additional chemotherapy, radiation therapy, targeted therapy or immunotherapy.
2. Known history of hypersensitivity to macromolecular protein preparation or any components of the SHR- 1210 formulation.
3. Subjects before or at the same time with other malignant tumors (except which has cured skin basal cell carcinoma and cervical carcinoma in situ);
4. Subjects with any active autoimmune disease or history of autoimmune disease
5. Uncontrolled clinically significant heart disease, including but not limited to the following: (1) > NYHA II congestive heart failure; (2) unstable angina, (3) myocardial infarction within the past 1 year; (4) clinically significant supraventricular arrhythmia or ventricular arrhythmia requirement for treatment or intervention;
6. Active infection or an unexplained fever > 38.5°C during screening or before the first scheduled day of dosing (subjects with tumor fever may be enrolled at the discretion of the investigator);
7. Received a live vaccine within 4 weeks of the first dose of study medication.
8. Pregnancy or breast feeding.
9. Decision of unsuitableness by principal investigator or physician-in-charge.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2017-07-19 (Actual); Primary Completion 2018-07-20 (Actual); Study Completion 2019-11-01 (Actual)

PRIMARY OUTCOMES:
Incidence of Treatment-Emergent Adverse Events | Through study completion, an average of half a year
  Adverse events (AE), Serious Adverse Event(SAE)

SECONDARY OUTCOMES:
ORR | Through study completion, an average of 1 year
  Objective Response Rate
PFS | 1year and 3years
  Progression-Free Survial
OS | 1year and 3years
  Overall Survival

CONTACTS AND LOCATIONS:
Overall Officials: PING WANG, MD.PHD, Principal Investigator — Tianjin Medical University Institute and Hospital
Locations (1):
- Department of Radiation Oncology, Tianjin Medical University Cancer Hospital, Tianjin, Tianjin Municipality, China

REFERENCES:
- [Derived] Wei H, Li Y, Guo Z, Ma X, Li Y, Wei X, Han D, Zhang T, Chen X, Yan C, Zhou J, Pang Q, Wang P, Zhang W. Comparison of dynamic changes in the peripheral CD8+ T cells function and differentiation in ESCC patients treated with radiotherapy combined with anti-PD-1 antibody or concurrent chemoradiotherapy. Front Immunol. 2022 Nov 21;13:1060695. doi: 10.3389/fimmu.2022.1060695. eCollection 2022. PMID 36479110